CLINICAL TRIAL: NCT04196699
Title: Evaluating the Feasibility, Acceptability and Pre Testing the Impact of a Self-management and Tele Monitoring Program for COPD Patients in Lebanon: Protocol for a Feasibility Study
Brief Title: Evaluating the Feasibility, Acceptability and Pre Testing the Impact of a Self-management and Tele Monitoring Program for COPD Patients in Lebanon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Paris 13 (Other)
Collaborators: Lebanese University (Other); Hotel Dieu Hospital (Other)
Responsible Party: Principal Investigator, Rita Nohra, Principal Investigator, University of Paris 13
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Feasibility study (Neith)
Record Dates: First submitted 2019-12-04; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Self-Management

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: self-management program — Our intervention will be based on the following framework and will consist of 3 phases :
  Phase I: At the end of a medical consultation, the doctor will offer the patient the opportunity to benefit from a nursing consultation and remote monitoring to better manage his COPD. A nursing consultation will be scheduled during which the nurse will explain the procedure, obtain the written consent of the patient, and develop an educational diagnosis with the participation of the patient.
  Phase II: During the next six weeks education sessions will be provide to the participants and a telephone number will be available in case of emergency and for any additional information.
  Phase III: A final consultation will be scheduled at the nurse office to evaluate the patient's achievements and modify his/her educational assessment. A telephone follow-up will be conducted after one month to assess the maintenance of learning.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) has a significant impact on quality of life and is costly to the health care system. It has been demonstrated that a self-management program improves quality of life, but programs are not universally available and telehealth interventions can provide home-based support, but have mixed results.

The aims of this study are to (1) assess the feasibility and acceptability of a 6 weeks' educational program related to self-management with remote monitoring for Lebanese COPD patients; (2) pre-test its impact on quality of life, emergency visits, and rate of rehospitalization, and (3) to make recommendations for a future randomized trial.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility, acceptability and pre-test the impact of a nursing consultation and tele-monitoring in Lebanon. It will be conducted at the Hôtel-Dieu de France (HDF) hospital, one of the largest university hospitals in Beirut, and will use quantitative and qualitative methods in pre- and post-intervention to collect data over a period of 3 months. Data will be collected by two researchers. A consent form will be signed by each participant prior to the intervention. Patients will be informed about the purpose of the study, the course of the intervention, and the freedom to withdraw from the study at any time. Their consent for the video recording will also be taken.

This study is the first to evaluate the application of telehealth to optimize COPD management in Lebanon. The results of this study will provide evidence regarding the efficacy and feasibility of this approach for Lebanese patients with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Adult,18 years of age or older
* Male or female
* Outpatient
* With moderate (GOLD 2) or severe (Gold 3) COPD.
* Cognitively capable, with an adequate health status to participate in the study according to the clinical consensus between nurses and physicians.

Exclusion Criteria:

* Patients diagnosed with lung cancer
* Patients who have cognitive problems related to memory loss or speech disorders that would not allow a constructive exchange

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2020-05-28 (Estimated); Study Completion 2020-06-28 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 2 month
  Based on "Pre-Referral intervention team inventory" we have created our own evaluation grid composed of 9 questions. Answers ranged between strongly agree to strongly disagree.
Adoption | 2 month
  Based on "adoption of information technology innovation" we have created our own evaluation grid composed of 5 questions. Patient must choose one of the proposed answers that best suits him/her.
Adequacy | 2 month
  Based on "Parenting strategies questionnaire" we have created our own qualitative evaluation grid composed of three questions. the patient must assign a score to each question that varies between 0 and 10.
Fidelity | 2 month
  Fidelity will be assessed by comparing the protocol of the intervention with what will be done in the field.
Cost | 2 month
  Based on "Utilization and Cost Questionnaire" we have created our own qualitative evaluation grid composed of 4 questions.
Coverage | 2 month
  Based on "levels of institutionalization". it is composed of 15 multiple-choice questions. Based on the average of the responses, the score will range from a low to high level of institutionalization.

SECONDARY OUTCOMES:
Impact on quality of life | 3 month
  We will use the COPD assessment test (CAT) to evaluate the quality of life of participants.
  CAT is composed of eight questions measured on a 5-point scale, with a score ranging from 0 to 40. Highest scores indicate a higher impact of COPD on patients' quality of life.
Rehospitalization rate | 3 month
  The hospital register of each participant will be consulted to collect and evaluate the number of hospitalizations during the year preceding the intervention and during the intervention
Emergency visit | 3 month
  The hospital register of each participant will be consulted to collect and evaluate the emergency room visits during the year preceding the intervention and during the intervention
Respiratory health status | 3 month
  COPD clinical questionnaire (CCQ). It consists of 10 questions in 3 domains (symptoms, functional state, and mental state). All scores ranged from 0 to 6, and the final score is the mean of the sum of all items, with a higher score indicating a lower health status.
Anxiety | 3 month
  "Hospital Anxiety and Depression" (HAD). It includes 14 rated items from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), resulting in two scores (maximum score of each score = 21).